CLINICAL TRIAL: NCT01386151
Title: Safety and Efficacy of Parenteral KGF in Moderate Asthmatic Subjects
Brief Title: A Study to Assess Safety and Efficacy of a Novel Treatment, Keratinocyte Growth Factor (KGF), in Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHM MED 0879
Record Dates: First submitted 2011-06-24; First posted 2011-06-30 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Bronchial Asthma
Keywords: Moderate asthmatic, uncontrolled
MeSH Terms: conditions — Asthma | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study drug (Active Comparator): Keratinocyte growth factor (KGF) will be administered intravenously in a 'collapsed dose' regime of 180ug/kg on day 0 and day 11.
  Interventions: Drug: Keratinocyte Growth factor
- Placebo (Placebo Comparator): Saline will be used as a placebo comparator
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Keratinocyte Growth factor — KGF will be administered intravenously in a 'collapsed dose' regime of 180ug/kg on day 0 and day 11
  Other Names: Palifermin, rhKGF, Kepivance
  Arms: Study drug
Drug: Saline placebo — Normal (0.9%) saline will be used as a placebo.
  Arms: Placebo

SUMMARY:
This study will look at the permeability, or 'leakiness' of the airway epithelium (the inner lining of the lung) in asthmatic patients. Increased leakiness of this lining has been shown in asthmatic patients by other studies, not only in the lung but also possibly in the gut, perhaps reflecting a widespread defect. This leakiness may underline the interaction between the environment and a person's genetic make up, and may contribute to why some people get asthma, and how severe it is. Increased leakiness may allow increased exposure to inhaled allergic substances, helping to perpetuate the inflammation in the lungs that is a hallmark of asthma.

Specifically, this study will attempt to modify and reduce this permeability through the use of a substance called 'keratinocyte growth factor', or 'kgf'. KGF is a naturally occuring human protein, which is involved in stimulating the growth of cells lining the layers of the skin and gut, helping to repair damage and maintain their structure. It has been manufactured in a laboratory as the commercial compound 'Palifermin', which has already been used in humans to reduce damage to the lining of the mouth after chemotherapy. The study will see if Palifermin can similarly improve the lining of the lung in asthma patients and improve their symptoms. To date no treatments have been used in this area in asthma, and if successful the study will open up a whole new area of therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years, either gender
* Confirmed diagnosis of asthma for > 1 year as defined by BTS guidelines, requiring treatment with high dose inhaled corticosteroids +/- long acting β2 agonists, with persisting symptoms requiring use of short-acting beta agonist therapy >3x/week.
* Never-smoker or ex-smoker, having stopped >1 year ago, with <10 pack year history.
* Subject must understand the procedures of the study and agree to participation in the study by providing written informed consent
* Subject considered fit enough to undergo lung function testing including provocation tests, and bronchoscopy.
* Subject must not be participating in another clinical trial or have done so within the last 12 weeks.

Exclusion Criteria:

* Patients requiring regular maintenance oral steroids for their asthma, or those who are adhering to symbicort SMART single inhaler regime.
* Pregnancy (where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test >5mIU/ml), an intention to become pregnant or breast-feeding (lactating).
* Subjects with active lung disease other than asthma
* Significant medical (cardiopulmonary, neurological, renal, endocrine, gastrointestinal, psychiatric, hepatic or haematological)co-morbidity which in the view of the investigator could impact on the interpretation of results or participation in the trial, or which is uncontrolled with standard treatment.
* Current participation in another clinical trial or previous participation within the last 12 weeks.
* Alcohol or active drug abuse.
* Ongoing allergen desensitisation therapy
* Regular use of sedatives, hypnotics, tranquilisers
* Cancer or previous history of cancer
* Inability to understand directions for dosing and study assessment.
* Inability to be contacted in case of emergency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in PD15 Mannitol | Baseline (7 days prior to drug), during drug administration period (3 days after first dose of drug), and short/intermediate term post drug period (3, 6 and 24 days after second drug administration)
  A standard bronchoprovocation test, the mannitol test, will be used to assess airway hyperreactivity (measured as the dose required to drop FEV1 (forced expiratory volume in 1 second) by 15%, PD15)

SECONDARY OUTCOMES:
Change in PC20 Metacholine | Baseline (6 days prior to drug) and short/intermediate term post drug period (7 and 25 days after second drug administration)
  A standard bronchoprovocation test, metacholine challenge, will be used to assess airway hyperreactivity (by measuring the concentration needed to drop FEV1 by 20%, PC20)
Change in asthma symptoms | ACQ is measured weekly during study. AQLQ is measured at baseline screening visit, and on day 35 (35 days post first administration of drug).
  Symptoms will be assessed using standardised questionnaires, Asthma control questionnaire (ACQ) and Asthma Quality of Life questionnaire (AQLQ)
Short acting beta-agonist use/PEFR variability | Throughout study
  A diary card will be used throughout the study for participants to record beta-agonist use and morning/evening peak expiratory flow rates (PEFR), from the latter PEFR variability will be calculated
Adverse event reporting | Throughout study
  Adverse events will be recorded if they occur
Epithelial integrity/activation | Specimens are taken at 2 bronchoscopies, the first before the drug (4 days prior to the first drug administration) and the second after the drug (21 days after the first drug administration)
  Bronchial biopsies, brush specimens and lavage fluid before and after intervention will be analysed to determine markers of activation, inflammation and epithelial integrity
Epithelial proliferation | Specimens are taken at 2 bronchoscopies, the first before the drug (4 days prior to the first drug administration) and the second after the drug (21 days after the first drug administration)
  Bronchial biopsy specimens will be analysed for markers of proliferation e.g. Ki67 before and after treatment
Exhaled nitric Oxide | This is measured on the same days as PD15 mannitol, with an additional baseline measurement at the screening visit
  Exhaled nitric oxide, as a surrogate marker of eosinophilic inflammation, will be measured before/during and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Howarth, BSc, MBBS, Principal Investigator — Reader in Medicine and Honorary Consultant Physician, Southampton General Hospital
Locations (1):
- Biomedical Research Unit (Respiratory), Southampton, Hampshire, United Kingdom